CLINICAL TRIAL: NCT02667847
Title: Preoperative Anxiety Evaluation: a New Visual Smileys Scale
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Corresponding Author, Cedars-Sinai Medical Center
Other Study IDs: Pro00030220
Record Dates: First submitted 2015-02-26; First posted 2016-01-29 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Anxiety, Preoperative
Keywords: preoperative anxiety assessment; levels of preoperative anxiety using two different scales
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preoperative patients: Preoperative patients were asked to verbally rate their anxiety 1=on a scale from 0-10 and 2=using the new smiley scale

SUMMARY:
Preoperative anxiety is a complex clinical concept with both physiological and psychological consequences.

DETAILED DESCRIPTION:
This study looks at the need for a more user friendly, rapid tool for measuring preoperative anxiety, specifically by evaluating the visual smileys scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* undergoing surgery at Cedars Sinai Medical Center

Exclusion Criteria:

* did not receive sedative or narcotic prior to the interview

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients undergoing surgery at Cedars Sinai Medical Center
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Anxiety level, as measured by verbal rating scale or visual smileys scale | up to 5 minutes
  in preoperative setting

SECONDARY OUTCOMES:
scale preference | up to 5 minutes
  in preoperative setting, comparing verbal rating scale and visual smileys scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States